CLINICAL TRIAL: NCT04365179
Title: An Open-Label Phase 1b Study of NEROFE, a Novel Hormone-Peptide in Adult Patients With Advanced Myelodysplastic Syndrome (MDS) and Acute Myelogenous Leukemia (AML)
Brief Title: Study of NEROFE, a Novel Hormone-Peptide in Adult Patients With Advanced MDS and AML
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Immune System Key Ltd (Industry)
Collaborators: University of Miami Sylvester Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20190675
Record Dates: First submitted 2020-04-12; First posted 2020-04-28 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Advanced MDS; AML
MeSH Terms: interventions — tumor-cells apoptosis factor, human

STUDY DESIGN:
Intervention Model Description: traditional 3+3 design
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NEROFE (Experimental): Dose Level - Nerofe Dose
  -1 - 6mg/m2
  1. - 12 mg/m2
  2. - 24 mg/m2
  3. - 48 mg/m2
  4. - 96 mg/m2
  5. - 150mg/m2
  Interventions: Drug: Nerofe

INTERVENTIONS:
Drug: Nerofe — Up to 12 cycles of 28 days are planned. If patients are deriving benefit, treatment may continue past 12 cycles.
  Cycle 1: During Cycle 1, assigned NEROFE doses will be administered by intravenous (IV) infusion over 1 hour on Days 1, 3, 5, 8, 10, 12, 15, 17, 19, 22, 24 and 26.
  Cycles 2-12: Subsequent cycles will be administered as above, presuming that patients do not meet criteria for study withdrawal during cycle 1.

SUMMARY:
This is an open-label Phase 1b study of NEROFE following a traditional 3+3 design to assess safety and to determine the Recommended Phase 2 Dose (RP2D) of NEROFE in patients with MDS or AML. IV NEROFE will be administered three times per week on alternate days. The exact dosage will be determined using the body surface area (BSA) measured on Day 1 of each cycle.

DETAILED DESCRIPTION:
NEROFE monotherapy may be administered for a maximum of 12 cycles provided that the patient tolerates treatment and there is evidence of clinical benefit. If patients are receiving clinical benefit, they may continue past 12 cycles.

Patients will be followed for a minimum of 30 days after the last dose of NEROFE monotherapy.

After this 30 day period, patients will only be followed for the resolution of any ongoing adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of one of the following:

   1. Relapsed/refractory Acute Myelogenous Leukemia (AML) where no alternative life prolonging therapy exists. Adverse genetic risk treatment naïve patients may also be considered eligible if, in the opinion of the investigator, these patients are unlikely to benefit from alternative therapy (e.g., an older patient with adverse risk MDS who progresses to AML after failing treatment for MDS (i.e. hypomethylating agent (HMA) or HMA and Venetoclax and is not a candidate for traditional AML induction chemotherapy).
   2. Relapsed/refractory Myelodysplastic Syndrome (MDS) those who fail to achieve a complete remission (CR) with at least 4 cycles of HMA (e.g. decitabine or azacitidine); or those who have progressive disease or have intolerance of HMA therapy after at least 2 cycles. Intolerance to HMA includes those patients forced to stop the HMA after at least 2 cycles due to severe infections/worsening cytopenias and are otherwise considered eligible. Patients with MDS have to have intermediate, high, or very high risk disease by International Prognostic Scoring System - Revised (IPSS-R score).
2. Adult male or female patients 18 years of age or older.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1 or 2.
4. Patients must satisfy the following laboratory criteria:

   1. Pre-treatment bone marrow staining must demonstrate expression of the ST2 receptor by IHC (low or high expression is allowed).
   2. Total bilirubin < 1.5 x greater upper limit of normal (UNL). Elevated indirect bilirubin associated with post-transfusion hemolysis is allowed.
   3. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) must be < 3 x UNL
   4. Creatinine < 2 x UNL or calculated creatinine clearance > 40 ml/min; or Estimated Glomerular Filtration Rate (eGFR) <50 according to MDRD (Modification of Diet in Renal Disease) method.
   5. White blood cell count (WBC) < 25,000/uL before the administration of NEROFE on Cycle 1 Day 1. Use of hydroxyurea to control the level of circulating leukemic blast cell counts is allowed before and during the study.
5. Suitable venous access to allow for all study related blood sampling (safety and research).
6. Estimated life expectancy, in the judgment of the investigator, which will permit receipt of at least 8 weeks of treatment.
7. Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without jeopardy to future medical care.
8. Female patients who are:

   1. Postmenopausal for at least one year before the screening visit, OR
   2. Surgically sterile, OR
   3. If they are of childbearing potential:

   Agree to practice one highly effective method and one additional effective (barrier) method of contraception, at the same time, form the time of signing the informed consent through 4 months after the last does of study drug (female and male condoms should not be used together), OR Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant. (Periodic abstinence e.g. calendar, ovulation, symptothermal, postovulation methods; withdrawal; spermicides only; and lactational amenorrhea are not acceptable methods of contraception).
9. Male patients even if surgically sterilized (e.g. status post vasectomy), who:

   1. Agree to practice effective barrier contraception during the entire study treatment period and through four months after the last dose of study drug (female and male condoms should not be used together), OR
   2. Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant. (Periodic abstinence e.g. calendar, ovulation, symptothermal, postovulation methods; withdrawal; spermicides only; and lactational amenorrhea are not acceptable methods of contraception).
10. Able to undergo bone marrow examination at screening

Exclusion Criteria:

1. Patients with a diagnosis of acute promyelocytic leukemia (APL).
2. Screening bone marrow slide without staining for ST2 receptor. (Low or High expression by Immunohistochemistry [IHC] allowed on study).
3. Therapy with any investigational products, anti-neoplastic therapy, or radiotherapy within 14 days of Cycle 1 Day 1. Patients actively receiving hydroxyurea are eligible and may continue to receive this medication during treatment on this protocol.
4. Candidates for standard and/or potentially curative treatments. (A candidate is defined as a patient that is both eligible and willing to have these treatments.)
5. Major surgery within 30 days of the first dose of any study drug or a scheduled surgery during study period.
6. Grade 2 or higher diarrhea (as defined by NCI CTCAE Version 5.0) despite optimal anti-diarrheal supportive care within 7 days prior to Cycle 1 Day 1.
7. Known cardiopulmonary disease as defined by one of the following:

   1. Clinically significant arrhythmia including: history of polymorphic ventricular fibrillation or torsade de pointes; atrial fibrillation > 7 days and requiring cardioversion in the 4 weeks before screening; incompletely controlled, symptomatic atrial fibrillation. Patients with Afib are permitted to enroll if it is < Grade 3 for a period of 6 months or greater and the rate is controlled with a stable regimen.
   2. Congestive heart failure (New York Heart Association (NYHA) Class III or IV; or Class II with a recent decompensation requiring hospitalization or referral to a heart failure clinic within four weeks of screening; myocardial infarction (MI) and/or revascularization (e.g.

      coronary bypass graft/stent) within 6 months of first dose of study drug.;
   3. Patients with ischemic heart disease who have had acute coronary syndrome (ACS), MI< and/or revascularization greater than 6 months before screening and who are without cardiac symptoms may enroll.
   4. Moderate to severe aortic and/or mitral valve stenosis or other ongoing valvulopathy;
   5. Pulmonary hypertension (symptomatic)
   6. Prolonged rate corrected QT (QTc) interval >480 msec, calculated according to institutional guidelines;
   7. Known, active left ventricular ejection fraction (LVEF) < 50% as assessed by echocardiogram or radionuclide angiography (not required at screening);
   8. Known moderate to severe chronic obstructive pulmonary disease (COPD), interstitial lung disease and/or pulmonary fibrosis (e.g., requiring home O2 therapy).
8. Active and uncontrolled infection or severe infectious disease, such as severe pneumonia, meningitis, or septicemia (stable or resolving infection on antibiotics is allowed).
9. Known human immunodeficiency virus (HIV) seropositive.
10. Known Hepatitis B surface antigen seropositive (note: patients who have isolated positive hepatitis B core antibody [e.g. in the setting of negative hepatitis B surface antigen and negative hepatitis B surface antibody] must have an undetectable hepatitis viral load).
11. Known or suspected active hepatitis C infection. Patients with treated Hep C treated with a negative viral load are eligible.
12. Females of child bearing potential who refuse to practice two effective methods of contraception at the same time or abstain from heterosexual intercourse from the time of signing consent through four months after the last dose of study drug.
13. Males of child bearing potential who refuse to practice effective barrier methods of contraception at the same time or abstain from heterosexual intercourse from the time of signing consent through four months after the last dose of study drug.
14. Female patients who are both lactating or breastfeeding, or have a positive serum pregnancy test during the screening period or a positive urine pregnancy test on Day 1 before the first dose of study drug.
15. Female patients who intend to donate eggs (ova) during the course of this study or within four months after receiving their last dose of study drug.
16. Male patients who intend to donate sperm during the course of this study or within four months after receiving their last dose of study drug.
17. Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of study procedures.
18. Symptomatic central nervous system (CNS) involvement.
19. Diagnosed or treated for another malignancy within 2 years with evidence of residual disease.
20. Known hepatic cirrhosis or severe pre-existing hepatic impairment.
21. Patients with uncontrolled coagulopathy or bleeding disorder.
22. Use of systemic steroids (prednisone) >10mg/day or any equivalent corticosteroids within 7 days of Cycle 1 Day 1. Patients on other immunosuppression (such as post-transplant) and also ineligible. Patients with active, uncontrolled GVHD (Graft Versus Host Disease) are also ineligible. Otherwise patients are eligible post-bone marrow transplantation.
23. Life-threatening illnesses unrelated to cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2020-06-18 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Assessing change in IWG (International Working Group) Criteria to evaluate response to Nerofe Treatment for MDS patients | At Screening (Day 1), at cycle 3 (Day 1) at cycle 5 (Day 1), at cycle 7 (Day 1), at cycle 9 (Day 1) at cycle 11 (Day 1) and at End of Treatment Visit. Cycle length is 28 days. Through study completion, an average of 1 year.
  Bone Marrow samples to measure percentage of blasts (%). Range 0-30% (the higher percentage the worse outcome)
Assessing change in IWG (International Working Group) Criteria to evaluate response to Nerofe Treatment for MDS patients. A calculation of several variables. | At every cycle on Day 1, Day 3, Day 8, Day 10, Day 12, D15, Day 17, Day 19, Day 22, Day 24, Day 26 and Day 28 (cycle length is 28 days), and at End of Treatment Visit, through study completion, an average of 1 year.
  Complete Blood Count (CBC) to measure hemoglobin (g/dL). Range 4-18 (4 worse outcome and 18 best outcome)
Assessing change in IWG (International Working Group) Criteria to evaluate response to Nerofe Treatment for MDS patients. A calculation of several variables. | At every cycle on Day 1, Day 3, Day 8, Day 10, Day 12, D15, Day 17, Day 19, Day 22, Day 24, Day 26 and Day 28 (cycle length is 28 days), and at End of Treatment Visit, through study completion, an average of 1 year.
  Complete Blood Count (CBC) to measure absolute neutrophil count (x10^9/L). Range 0-15 (the higher the score the better outcome).
Assessing change in IWG (International Working Group) Criteria to evaluate response to Nerofe Treatment for MDS patients. A calculation of several variables. | At every cycle on Day 1, Day 3, Day 8, Day 10, Day 12, D15, Day 17, Day 19, Day 22, Day 24, Day 26 and Day 28 (cycle length is 28 days), and at End of Treatment Visit, through study completion, an average of 1 year.
  Complete Blood Count (CBC) to measure platelets (x10^9/L). Range 0-2000 (the higher the score the better outcome).
Assessing change in IWG (International Working Group) Criteria to evaluate response to Nerofe Treatment for MDS patients. A calculation of several variables. | At every cycle on Day 1, Day 3, Day 8, Day 10, Day 12, D15, Day 17, Day 19, Day 22, Day 24, Day 26 and Day 28 (cycle length is 28 days), and at End of Treatment Visit, through study completion, an average of 1 year.
  Complete Blood Count (CBC) to measure cytogenetic abnormalities. Range from very good (0) to very poor (4).
Assessing change in ELN 2017 (European Leukemia Net) Criteria to evaluate response to Nerofe Treatment for AML patients | At Screening (Day 1), at cycle 3 (Day 1) at cycle 5 (Day 1), at cycle 7 (Day 1), at cycle 9 (Day 1) at cycle 11 (Day 1) and at End of Treatment Visit. Cycle length is 28 days. Through study completion, an average of 1 year.
  Bone Marrow samples to measure percentage of blasts (%). Range 0-30% (the higher percentage the worse outcome)
Assessing change in ELN 2017 (European Leukemia Net) Criteria to evaluate response to Nerofe Treatment for AML patients. A calculation of several variables. | At every cycle on Day 1, Day 3, Day 8, Day 10, Day 12, D15, Day 17, Day 19, Day 22, Day 24, Day 26 and Day 28 (cycle length is 28 days), and at End of Treatment Visit, through study completion, an average of 1 year.
  Complete Blood Count (CBC) to measure absolute neutrophil count (x10^9/L). Range 0-15 (the higher the score the better outcome)
Assessing change in ELN 2017 (European Leukemia Net) Criteria to evaluate response to Nerofe Treatment for AML patients. A calculation of several variables. | At every cycle on Day 1, Day 3, Day 8, Day 10, Day 12, D15, Day 17, Day 19, Day 22, Day 24, Day 26 and Day 28 (cycle length is 28 days), and at End of Treatment Visit, through study completion, an average of 1 year.
  Complete Blood Count (CBC) to to measure platelets (x10^9/L). Range 0-2000 (the higher the score the better outcome).
Assessing change in ELN 2017 (European Leukemia Net) Criteria to evaluate response to Nerofe Treatment for AML patients. A calculation of several variables. | At every cycle on Day 1, Day 3, Day 8, Day 10, Day 12, D15, Day 17, Day 19, Day 22, Day 24, Day 26 and Day 28 (cycle length is 28 days), and at End of Treatment Visit, through study completion, an average of 1 year.
  Complete Blood Count (CBC) to measure cytogenetic abnormalities. Range from very good (0) to very poor (4).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Miami Hospital and Clinics / Sylvester Comprehensive Cancer Center, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No